CLINICAL TRIAL: NCT02795442
Title: Daily Protein Intake Patterns on Energy Metabolism and the Motivation to Snack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GFHNRC500
Record Dates: First submitted 2016-06-06; First posted 2016-06-10 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Even protein (Experimental): Menu to provide 90 g of protein per day in an even distribution of 30 g at each meal.
  Interventions: Other: Even protein
- Skewed protein (Experimental): Menu to provide 90 g of protein per day in a skewed distribution of 10 g at breakfast, 15 g at lunch and 65 g at dinner.
  Interventions: Other: Skewed protein

INTERVENTIONS:
Other: Even protein — 5 day intake of even protein 3 day rotating menu.
  Arms: Even protein
Other: Skewed protein — 5 day intake of skewed protein 3 day rotating menu.
  Arms: Skewed protein

SUMMARY:
The purpose of this study is to determine if when one eats protein can change how the body uses food for energy. Researchers will also test if eating a high protein breakfast can change one's craving for snack foods.

DETAILED DESCRIPTION:
The purpose of this study is to determine if consuming 30 g of high-quality protein at each meal can increase fat utilization and shift between-meal snack choices. While the benefits of high-protein diets are well known, little is known about the optimal amount of protein that should be eaten at each meal. Most Americans eat little protein at breakfast and lunch and most of their protein at the evening meal. Current guidelines for protein are based on body weight; however, recent evidence indicates that absolute amounts of protein at each meal are needed to maintain metabolically active fat-free mass. This suggests that a more even protein consumption pattern across daily meals may positively influence energy metabolism. In addition, recent evidence indicates that protein may reduce activity in the food reward areas of the brain. This suggests that protein may influence between-meal snacking by decreasing the relative reinforcing value (RRV) of highly rewarding snack foods. The RRV of a food is an empirical measure of its motivating value and energy-dense foods are highly reinforcing, especially for obese individuals. This study will be the first to investigate the role of the daily distribution of protein intake on energy metabolism and modifying snacking behavior.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 25 kg/m2
* BMI ≥ 30 kg/m2 but < 34.5 kg/m2
* able to understand and sign the informed consent
* able to provide own transportation to the Center
* free of any major illness/disease
* usual protein intake within the acceptable macronutrient distribution range (10 to 30%)
* constant habitual activity patterns within the last 3 months
* females of childbearing age must be on birth control for a minimum of 3 months prior to study start and have regular menstrual cycles

Exclusion Criteria:

* unable or unwilling to consume animal products
* have had more than a 10% change in body weight within the past 2 months
* are participating in a weight loss diet/exercise program
* are consuming a specialized diet
* currently or planning on becoming pregnant during the study timeline
* lactating
* have a metabolic illness/disease
* have uncontrolled hypertension
* have ever had cancer
* have an infectious disease
* suffer from alcohol or drug abuse
* use tobacco and e-cigarette products on a regular basis
* have the presence of acute illness
* taking medications known to affect energy expenditure and appetite

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Fat, carbohydrate, and protein utilization | 4 hours after meal consumption
  The effect of consuming two patterns of daily protein intake on the use of fat, carbohydrate and protein for energy.
Relative reinforcing value (RRV) of energy-dense snack foods | 2 hours after breakfast consumption
  The effect of consuming a high-protein or a low-protein breakfast on the RRV of energy-dense snack foods to a healthy snack food alternative.

SECONDARY OUTCOMES:
Peripheral neurotransmitter metabolites | 2 hours
  The effect of consuming a high-protein or low-protein breakfast and an energy-dense snack food on dopamine and serotonin metabolite plasma concentrations.
Psychoactive Effect Questionnaire | 2 hours
  The effect of consuming a high-protein or low-protein breakfast and an energy-dense snack food on the number of positive responses on the Psychoactive Effects Questionnaire.
Satiety visual analog scales | 4 hours after meal consumption
  The effect of consuming two patterns of daily protein intake on subjective measures of satiety.

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT02795442/ICF_000.pdf